CLINICAL TRIAL: NCT02441322
Title: High Resolution MRI and MRS to Evaluate Therapeutic Response to Novo-TTF in Newly and Recurrent Glioblastomas
Brief Title: Evaluating Therapeutic Response to Novo-TTF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 12314; 820817 (Other: IRB)
Record Dates: First submitted 2015-02-11; First posted 2015-05-12 (Estimated); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Glioblastoma Multiforme
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Methods to identify treatment response (Experimental): The investigators will study how well these advanced MRI methods are in accurately identifying response to Novo-TTF in comparison to standard MRI methods for evaluation of treatment response. Using advanced MRI imaging techniques may help assess treatment response earlier than changes in tumor volume which can be measured with standard MRI methods.
  Interventions: Device: Novo-TTF

INTERVENTIONS:
Device: Novo-TTF — Procedures: MRI and advanced MRI sequence Advanced brain MRI's with special sequences will be obtained. First MRI prior to starting Novo-TTF therapy, second MRI up to 2-3 weeks after beginning therapy, third MRI up to 2 months from starting treatment and the last MRI up to 4 months after starting treatment.
  Other Names: Optune

SUMMARY:
This study is to assess the utility of high resolution 3D echo planar magnetic resonance spectroscopy (3D EPSI) in monitoring Novo-TTF response in glioblastoma multiforme (GBM) patients.

DETAILED DESCRIPTION:
The patient is being asked to have 4 MRI scans of their brain over the course of 6 months. Each MRI scan will take approximately 1 hour to complete. The first MRI scan will be performed once the patient is enrolled in the Novo-TTF treatment therapy, but prior to the initiation of Novo-TTF therapy. The second MRI scan will be performed up to 2-3 weeks after therapy had begun. The third MRI scan will be performed up to 2 months from the start of Novo-TTF treatment and the last MRI scan will be performed up to 4 months from the start of Novo-TTF treatment.

The MRI scans will be ordered by the principal investigator of the study and this will include standard MR imaging sequences along with advanced MR spectroscopy (MRS) to help identify response to Optune therapy. Please note: the only portion of the MRI scan that will be research-related are the MRS sequences. The other portion of the imaging will be considered as a standard of care MRI scan that will be reviewed by an attending physician, who will generate an MRI report in the electronic medical record system (EMS). The data collected from the advanced MRS sequences will be reviewed by the principal investigator and will be billed to the research study (you will be billed for the clinical MRI scan as a part of your standard of care).

The MRI study will be conducted at the Center for Advanced Magnetic Resonance Imaging and Spectroscopy in the Department of Radiology, University of Pennsylvania Medical Center. The study scans will be very similar to routine clinical MRI scans of the brain.

The patient will be asked to lie on a specially designed bed and a circular antenna will be placed around the patients head. The patient will be given earplugs to wear to decrease the banging noise caused by the imaging process. The earplugs do not block out all sound since the MRI tech's wish to stay in communication with the patient at all times. The MRI techs will then move the patient into the magnet, a large hollow cylinder, until the patients head is at the center. The study will then proceed. The MRI operator will inform the patient of the progress of the study. The patient will need to keep perfectly still during the scanning.

During each MRI scan, the patient will have an intravenous line (IV line) placed. The IV line allows the contrast agent to be injected into the patient's vein. MRI contrast agents are chemicals that travel through the bloodstream. They act like dyes to make MRI pictures brighter and easier to read.

When the study is complete, the patient will be moved out of the magnet. The MRI operator will ask that the patient please get up slowly since the patient has been lying still for a relatively long period of time.

The investigators will also review the patient's medical records for information about medical history, current and past medications and therapies, and other information related to the patient's GBM.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed or recurrent GBMs
* Received maximal debulking surgery and radiotherapy (protons or photons) concomitant with Temozolomide (40-75Gy)
* Patients may enroll in the study if received Gliadel wafers before entering the trial.
* Minimal dose for concomitant radiotherapy is 40 Gy
* Karnofsky scale of 60 or greater
* Life expectancy at least 3 months
* Must sign written informed consent
* Treatment start date at least 4 weeks out from surgery or as soon as skin healing/radiation reaction allows
* Measurable enhancing neoplasm on post contrast T1 weighted images and/or non enhancing FLAIR signal abnormality

Exclusion Criteria:

* Actively participating in another clinical treatment trial
* Pregnant
* Significant co-morbidities at baseline which would prevent maintenance Temozolomide treatment:

  1. Thrombocytopenia (platelet count less than 100 x 1000 per microlitre)
  2. Neutropenia (absolute neutrophil count less than 1.5 x 1000 per microlitre)
  3. CTC grade 4 non-hematological Toxicity (except for alopecia, nausea, vomiting)
  4. Significant liver function impairment AST or ALT 3 times the upper limit of normal
  5. Total bilirubin upper limit of normal
  6. Significant renal impairment (serum creatinine greater than 1.7 mg/dL)
* Implanted pacemaker, programmable shunts, defibrillator, deep brain stimulator, other implanted electronic devices in the brain, or documented clinically significant arrhythmias
* Infra-tentorial tumor
* Evidence of increased intracranial pressure (midline shift 5mm, clinically significant papilledema, vomiting and nausea or reduced level of consciousness)
* History of hypersensitivity reaction to Temozolomide or a history of hypersensitivity to DTIC.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-12; Primary Completion 2023-06 (Actual); Study Completion 2023-12 (Actual)

PRIMARY OUTCOMES:
Radiological response using standard of care bi monthly MRI scans | up to 2 years
  MRI scans will be used to help track radiological response to Optune therapy

SECONDARY OUTCOMES:
Overall survival (OS) | up to 2 years
  Evaluating patient overall survival on Optune therapy
Progression free survival time | up to 2 years
  Monitoring patient progression free survival time on Optune therapy
Treatment Response using modified RANO criterion | up to 2 years
  Optune therapy treatment response will be measured using modified RANO criterion

CONTACTS AND LOCATIONS:
Overall Officials: Suyash Mohan, Dr., Principal Investigator — University of Pennsylvania
Locations (1):
- University Of Pennsylvania, Philadelphia, Pennsylvania, United States